CLINICAL TRIAL: NCT03833167
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate Pembrolizumab Versus Placebo as Adjuvant Therapy Following Surgery and Radiation in Participants With High-risk Locally Advanced Cutaneous Squamous Cell Carcinoma (LA cSCC) (KEYNOTE-630)
Brief Title: Pembrolizumab (MK-3475) Versus Placebo Following Surgery and Radiation in Participants With Locally Advanced Cutaneous Squamous Cell Carcinoma (MK-3475-630/KEYNOTE-630)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-630; MK-3475-630 (Other: MSD); KEYNOTE-630 (Other: MSD); 2022-500395-57-00 (Registry Identifier: EU CT); U1111-1275-8212 (Registry Identifier: UTN); 2018-001974-76 (EudraCT Number)
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Squamous Cell
Keywords: Programmed Cell Death-1 (PD-1); Programmed Cell Death 1; PD1; Programmed Cell Death Ligand 1 (PD-L1); Programmed Cell Death Ligand 2 (PD-L2); PDL1; PDL2
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants receive 400 mg pembrolizumab by intravenous (IV) infusion administered on Day 1 of each 42-day cycle (Q6W) for up to 9 cycles. Participants that complete 9 cycles of pembrolizumab and experience biopsy-proven-disease recurrence may be eligible to receive up to 18 additional cycles of pembrolizumab in an open-label design.
  Interventions: Biological: Pembrolizumab
- Placebo (Placebo Comparator): Participants receive placebo by IV infusion administered on Day 1 of each 42-day cycle (Q6W) for up to 9 cycles. Participants treated with placebo who experience biopsy-proven-disease recurrence may be eligible to receive up to 18 cycles of pembrolizumab in an open-label design.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Pembrolizumab — 400 mg IV infusion
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab
Drug: Placebo — Placebo-matched IV infusion
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, study that compares pembrolizumab (MK-3475) with placebo given as adjuvant therapy in participants with high-risk locally advanced cutaneous squamous cell carcinoma (LA cSCC) that have undergone surgery with curative intent in combination with radiotherapy. The primary hypothesis is that pembrolizumab is superior to placebo in increasing recurrence free survival (RFS).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria include, but are not limited to:

* Has histologically confirmed cutaneous squamous cell carcinoma (cSCC) as the primary site of malignancy (metastatic skin involvement from another type of primary cancer or from an unknown primary cancer is not permitted)
* Has histologically confirmed locally advanced cutaneous squamous cell carcinoma (LA cSCC) with ≥1 high-risk feature(s) as the primary site of malignancy
* Has undergone complete macroscopic resection of all known cSCC disease with or without microscopic positive margins. For those participants with residual microscopic positive margin involvement, confirmation that additional re-excision is not possible must be provided
* Has completed adjuvant radiotherapy (RT) for LA cSCC with last dose of RT ≥4 weeks and ≤16 weeks from randomization
* Has received an adequate post-op dose of RT (either hypofractionated or conventional)
* Is disease free as assessed by the investigator with complete radiographic staging assessment ≤28 days from randomization
* Is not pregnant or breastfeeding
* Is not a person of childbearing potential (POCBP)
* Has a negative pregnancy test ≤72 hours before the first dose of study intervention.
* Has provided an archival or newly-obtained tumor tissue sample adequate for Programmed Cell Death Ligand 1 (PD-L1) testing as determined by central laboratory testing
* Has a life expectancy of >3 months
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 ≤10 days prior to the first dose of study intervention.

Exclusion Criteria:

Exclusion criteria include, but are not limited to:

* Has macroscopic residual cSCC after surgery and/or recurrence with active cSCC disease before randomization
* Has any other histologic type of skin cancer other than invasive cSCC (eg, basal cell carcinoma) that has not been definitively treated with surgery or radiation; Bowen's disease; Merkel cell carcinoma; or melanoma
* Has received prior therapy with an anti-programmed cell death receptor 1(PD-1), anti-PD-L1, or anti-programmed cell death receptor ligand 2 (PD-L2) agent or with an agent directed to another costimulatory or coinhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, CD137)
* Has received prior systemic anticancer therapy including investigational agents for cSCC ≤4 weeks prior to before start of study intervention.
* Has not recovered from all radiation-related toxicities and has not had radiation pneumonitis
* Has received a live vaccine ≤30 days prior to the first dose of study intervention
* Has received an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded. Other exceptions may be considered with Sponsor consultation. Note: Participants with low risk early-stage prostate cancer defined as below are not excluded: Stage T1c or T2a with a Gleason score ≤6 and a prostate-specific antigen (≤10 ng/ml) either treated with definitive intent or untreated in active surveillance that has been stable for the past year prior to study allocation. Early stage asymptomatic CLL without prior treatment and without any of the risk features (unmutated IGHV, lymphocytes >15,000μL, palpable lymph nodes) will be eligible for the study
* Has an active autoimmune disease that has required systemic treatment in past 2 years except replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid).
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (HCV; defined as HCV RNA [qualitative] is detected) infection
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study intervention
* Has had an allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2026-01-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (181):
- United States (30):
  - University of South Alabama, Mitchell Cancer Institute ( Site 1562), Mobile, Alabama
  - City of Hope Medical Center ( Site 1505), Duarte, California
  - UCSD Moores Cancer Center ( Site 1561), La Jolla, California
  - UCLA Hematology/Oncology - Westwood (Building 100) ( Site 1568), Los Angeles, California
  - University of California Davis Comprehensive Cancer Center ( Site 1560), Sacramento, California
  - Stanford University Medical Center ( Site 1503), Stanford, California
  - University of Colorado Cancer Center ( Site 1506), Aurora, Colorado
  - Smilow Cancer Center at Yale-New Haven ( Site 1507), New Haven, Connecticut
  - Boca Raton Regional Hospital ( Site 1551), Boca Raton, Florida
  - UF Health ( Site 1511), Gainesville, Florida
  - University of Miami Hospital and Clinics, Sylvester Cancer Center ( Site 1544), Miami, Florida
  - Winship Cancer Institute of Emory University ( Site 1512), Atlanta, Georgia
  - Indiana University Melvin and Bren Simon Cancer Center ( Site 1515), Indianapolis, Indiana
  - University of Iowa Hospital and Clinics ( Site 1514), Iowa City, Iowa
  - University of Kentucky School of Medicine & Hospitals ( Site 1542), Lexington, Kentucky
  - Massachusetts General Hospital ( Site 1518), Boston, Massachusetts
  - Dana Farber Cancer Center ( Site 1519), Boston, Massachusetts
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 1526), Hackensack, New Jersey
  - Northwell Health/ RJ Zuckerberg Cancer Center-Medical Oncology ( Site 1565), Lake Success, New York
  - Icahn School of Medicine at Mount Sinai ( Site 1575), New York, New York
  - Cleveland Clinic ( Site 1541), Cleveland, Ohio
  - Providence Portland Medical Center ( Site 1530), Portland, Oregon
  - UPMC Hillman Cancer Center ( Site 1570), Pittsburgh, Pennsylvania
  - MUSC Hollings Cancer Center ( Site 1533), Charleston, South Carolina
  - West Cancer Center - East Campus ( Site 1535), Germantown, Tennessee
  - Vanderbilt Ingram Cancer Center ( Site 1543), Nashville, Tennessee
  - The University of Texas-MD Anderson Cancer Center ( Site 1536), Houston, Texas
  - Huntsman Cancer Institute ( Site 1537), Salt Lake City, Utah
  - Inova Schar Cancer Institute ( Site 1538), Fairfax, Virginia
  - West Virginia University ( Site 1569), Morgantown, West Virginia
- Argentina (9):
  - Centro de Investigaciones Metabólicas (CINME)-Oncology ( Site 0028), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Centro Medico Privado CEMAIC ( Site 0024), Capital, Córdoba Province
  - Fundacion Estudios Clinicos-Oncology ( Site 0026), Rosario, Santa Fe Province
  - Centro Oncológico de Rosario ( Site 0003), Rosario, Santa Fe Province
  - Hospital Italiano- Sociedad Italiana de Beneficencia en Buenos Aires ( Site 0009), Buenos Aires
  - CEMIC ( Site 0012), Buenos Aires
  - Fundacion CIDEA ( Site 0001), CABA
  - Centro Oncologico Riojano Integral ( Site 0002), La Rioja
  - Centro Oncologico Norte ( Site 0023), Santiago del Estero
- Australia (7):
  - Chris OBrien Lifehouse ( Site 0051), Camperdown, New South Wales
  - Lismore Base Hospital ( Site 0050), Lismore, New South Wales
  - Orange Health Services ( Site 0053), Orange, New South Wales
  - Royal North Shore Hospital ( Site 0052), St Leonards, New South Wales
  - Gold Coast University Hospital ( Site 0054), Southport, Queensland
  - Sunshine Coast University Private Hospital-Coastal Cancer Care ( Site 0056), Sunshine Coast, Queensland
  - Alfred Health ( Site 0055), Melbourne, Victoria
- Brazil (8):
  - Oncocentro Ceara ( Site 0108), Fortaleza, Ceará
  - Hospital Erasto Gaertner ( Site 0101), Curitiba, Paraná
  - Hospital Tacchini ( Site 0111), Bento Gonçalves, Rio Grande do Sul
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia ( Site 0100), Ijuí, Rio Grande do Sul
  - Hospital Bruno Born ( Site 0107), Lajeado, Rio Grande do Sul
  - Hospital Sao Vicente de Paulo ( Site 0105), Passo Fundo, Rio Grande do Sul
  - Instituto Nacional de Câncer José Alencar Gomes da Silva - INCA-Pesquisa Clinica HC II ( Site 0103), Rio de Janeiro
  - A. C. Camargo Cancer Center ( Site 0116), São Paulo
- Canada (6):
  - Tom Baker Cancer Center ( Site 0161), Calgary, Alberta
  - Cross Cancer Institute ( Site 0159), Edmonton, Alberta
  - Juravinski Cancer Center ( Site 0151), Hamilton, Ontario
  - The Ottawa Hospital Cancer Centre ( Site 0154), Ottawa, Ontario
  - CIUSSS de l'Est-de-l'Île-de-Montréal ( Site 0163), Montreal, Quebec
  - McGill University Health Centre ( Site 0162), Montreal, Quebec
- Chile (4):
  - Enroll SpA ( Site 1654), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 1651), Santiago, Region M. de Santiago
  - James Lind Centro de Investigación del Cáncer ( Site 1653), Temuco, Región de la Araucanía
  - Bradford Hill Norte ( Site 1652), Antofagasta
- Colombia (6):
  - Sociedad de Cirugía de Bogotá - Hospital de San Jose ( Site 0201), Bogotá, Bogota D.C.
  - Instituto Nacional de Cancerologia E.S.E ( Site 0204), Bogotá, Bogota D.C.
  - Oncomedica S.A. ( Site 0205), Montería, Departamento de Córdoba
  - Oncologos del Occidente S.A. ( Site 0206), Pereira, Risaralda Department
  - Fundación Cardiovascular de Colombia ( Site 0207), Piedecuesta, Santander Department
  - Fundación Valle del Lili ( Site 0202), Cali, Valle del Cauca Department
- France (17):
  - Hopital ARCHET 2 ( Site 0356), Nice, Alpes-Maritimes
  - Hopital Saint Joseph ( Site 0376), Marseille, Bouches-du-Rhone
  - Hopital La Timone ( Site 0353), Marseille, Bouches-du-Rhone
  - Centre Hospitalier Universitaire de Caen Normandie-DERMATOLOGY ( Site 0365), Caen, Calvados
  - CHU Besancon - Hopital Jean Minjoz ( Site 0359), Besançon, Doubs
  - Centre Hospitalier de Valence ( Site 0377), Valence, Drome
  - C.H.U. de Nimes. Hopital Caremeau ( Site 0368), Nîmes, Gard
  - CHU de Bordeaux- Hopital Saint Andre ( Site 0370), Bordeaux, Gironde
  - Institut Claudius Regaud IUCT Oncopole ( Site 0354), Toulouse, Haute-Garonne
  - Centre Hospitalier Annecy Genevois ( Site 0361), Pringy, Haute-Savoie
  - CHU Montpellier. ( Site 0367), Montpellier, Herault
  - CHRU de Lille - Hopital Claude Huriez ( Site 0355), Lille, Nord
  - CHU Estaing ( Site 0360), Clermont-Ferrand, Puy-de-Dome
  - CH Lyon Sud Hospices Civils de Lyon ( Site 0350), Pierre-Bénite, Rhone
  - Hopital Avicenne ( Site 0358), Bobigny, Seine-Saint-Denis
  - Institut Gustave Roussy ( Site 0352), Villejuif, Val-de-Marne
  - CHU Poitiers ( Site 0375), Poitiers, Vienne
- Germany (8):
  - Universitaetsklinikum Tuebingen ( Site 0409), Tübingen, Baden-Wurttemberg
  - Klinikum Nürnberg Nord ( Site 0415), Nuremberg, Bavaria
  - Universitatsklinikum Giessen und Marburg GmbH ( Site 0413), Marburg, Hesse
  - Elbe Kliniken Stade-Buxtehude, Klinikum Buxtehude-Dermatologisches Zentrum ( Site 0411), Buxtehude, Lower Saxony
  - Medizinische Hochschule Hannover ( Site 0405), Hanover, Lower Saxony
  - Universitaetsklinikum Essen ( Site 0403), Essen, North Rhine-Westphalia
  - Universitaetsklinikum Berlin - Charite - Campus Mitte ( Site 0400), Berlin
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 0414), Hamburg
- Greece (5):
  - Andreas Syggros Hospital ( Site 0450), Athens, Achaia
  - Attikon University General Hospital of Athens ( Site 0454), Chaïdári, Attica
  - Metropolitan Hospital ( Site 0453), Neo Faliro, Attica
  - Papageorgiou General Hospital ( Site 0451), Thessaloniki
  - European Interbalkan Medical Center ( Site 0455), Thessaloniki
- Hungary (6):
  - Pecsi Tudomanyegyetem AOK ( Site 0501), Pécs, Baranya
  - Szegedi Tudomanyegyetem ( Site 0504), Szeged, Csongrád megye
  - Szabolcs Szatmar Bereg Megyei Korhazak es Egyetemi Oktatokorhaz ( Site 0500), Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Debreceni Egyetem. ( Site 0506), Debrecen, Vas County
  - Semmelweis Egyetem ( Site 0507), Budapest
  - Szent Imre Egyetemi Oktatokorhaz ( Site 0502), Budapest
- St. James s Hospital ( Site 1601), Dublin, Dublin, Ireland
- Israel (7):
  - Soroka University Medical Center ( Site 0555), Beersheba
  - Rambam Health Care Campus-Oncology Division ( Site 0552), Haifa
  - Haddassah Medical Organization - Ein Kerem ( Site 0553), Jerusalem
  - Meir Medical Center ( Site 0556), Kfar Saba
  - Rabin Medical Center ( Site 0550), Petah Tikva
  - Chaim Sheba Medical Center ( Site 0551), Ramat Gan
  - Sourasky Medical Center ( Site 0554), Tel Aviv
- Italy (5):
  - Instituto Tumori Giovanni Paolo II ( Site 0604), Bari, Apulia
  - Azienda Ospedaliero Universitaria Pisana ( Site 0603), Pisa, Tuscany
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 0600), Milan
  - Istituto Europeo di Oncologia ( Site 0602), Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 0601), Napoli
- Mexico (9):
  - San Lucas Cardiologica del Sureste S.A de C.V. ( Site 0722), Tuxtla Gutiérrez, Chiapas
  - Cimab SA de CV ( Site 0708), Torreón, Coahuila
  - Centro de Investigación Clínica de Alta Especialidad ( Site 0715), Torreón, Coahuila
  - Onco-Hematologia de Occidente ( Site 0716), Guadalajara, Jalisco
  - Hospital de Especialidades Centro Medico de Occidente ( Site 0704), Guadalajara, Jalisco
  - Consultorios de Medicina Especializada del Sector Privado ( Site 0701), Guadalajara, Jalisco
  - Centro de atencion e investigacion clinica en oncologia ( Site 0706), Mérida, Yucatán
  - Centro Estatal de Cancerologia de Chihuahua ( Site 0703), Chihuahua City
  - FAICIC Clinical Research ( Site 0700), Veracruz
- New Zealand Clinical Research (Auckland) ( Site 0800), Auckland, New Zealand
- Norway (3):
  - Haukeland sykehus ( Site 0851), Bergen, Hordaland
  - St. Olavs Hospital HF ( Site 0852), Trondheim, Sor-Trondelag
  - Oslo Universitetssykehus Radiumhospitalet ( Site 0850), Oslo
- Poland (4):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Oddzial w Krakowie ( Site 0959), Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 0951), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Chirurgii Onkologicznej, Transplantacyjnej i Ogólnej ( Site, Gdansk, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 0958), Gliwice, Silesian Voivodeship
- Portugal (5):
  - Hospital Particular do Algarve ( Site 1005), Faro
  - Instituto Portugues de Oncologia de Lisboa ( Site 1003), Lisbon
  - Hospital CUF - Tejo ( Site 1004), Lisbon
  - CHLN Hospital Santa Maria ( Site 1001), Lisbon
  - Inst. Portugues de Oncologia de Porto Francisco Gentil EPE ( Site 1000), Porto
- Romania (10):
  - S C Pelican Impex SRL ( Site 1108), Oradea, Bihor County
  - Hifu Terramed Conformal SRL ( Site 1111), Bucharest, București
  - Cardiomed SRL Cluj-Napoca ( Site 1104), Cluj-Napoca, Cluj
  - Institutul Oncologic Prof.Dr. Ion Chiricuta Cluj-Napoca ( Site 1113), Cluj-Napoca, Cluj
  - Spitalul Universitar CF Cluj-Napoca ( Site 1103), Cluj-Napoca, Cluj
  - S.C. Centrul de Oncologie Sf. Nectarie SRL ( Site 1101), Craiova, Dolj
  - S C Oncocenter Oncologie Medicala S R L ( Site 1106), Timișoara, Timiș County
  - Policlinica Oncomed SRL ( Site 1105), Timișoara, Timiș County
  - S.C.Focus Lab Plus S.R.L ( Site 1107), Bucharest
  - Spitalul de Psihiatrie Titan Dr. Constantin Gorgos ( Site 1112), Bucharest
- Russia (12):
  - Altay Regional Oncology Dispensary ( Site 1168), WBarnaularsaw, Altayskiy Kray
  - GBUZ Republican Clinical Oncological Dispensary-Antitumor drug therapy department ( Site 1171), Ufa, Baskortostan, Respublika
  - A. Tsyb Medical Radiological Research Center - branch of the National Medical Research Radiological, Obninsk, Kaluzskaja Oblast
  - Oncological Dispensary #2 of Ministry of Health of Krasnodar region ( Site 1159), Sochi, Krasnodarskiy Kray
  - N.N. Blokhin NMRCO ( Site 1153), Moscow, Moscow
  - FSCC FMBA of Russia ( Site 1163), Moscow, Moscow
  - First Moscow State Medical University n.a. I.M.Sechenov ( Site 1164), Moscow, Moscow
  - Hadassah Medical-Oncology department ( Site 1173), Moscow, Moscow Oblast
  - Nizhniy Novgorod regional clinical oncological dispensary ( Site 1169), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Railway Hospital of OJSC ( Site 1161), Saint Petersburg, Sankt-Peterburg
  - Udmurtia Republic Regional Clinical Oncology Dispensary ( Site 1158), Izhevsk, Udmurtiya Republic
  - Yaroslavl Regional SBIH Clinical Oncology Hospital ( Site 1152), Yaroslavl, Yaroslavl Oblast
- Spain (7):
  - Hospital Duran i Reynals ( Site 1254), Hospitalet Del Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla ( Site 1256), Santander, Cantabria
  - Hospital Clinic i Provincial Barcelona ( Site 1253), Barcelona, Catalonia
  - Onkologikoa - Instituto Oncologico de San Sebastian ( Site 1258), Doniostia - San Sebastian, Gipuzkoa
  - Hospital General Universitari Vall d Hebron ( Site 1252), Barcelona
  - Hospital Universitario Ramon y Cajal ( Site 1251), Madrid
  - Hospital Universitario Carlos Haya ( Site 1255), Málaga
- Ukraine (5):
  - Communal Non-Commercial Enterprise "Prykarpatski Clinical On-Department for daily treated patient (, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Institute of General and Emergency Surgery named after V.T. Zaitsev NAMS of Ukraine ( Site 1450), Kharkiv, Kharkivs’ka Oblast’
  - Limited Liability Company Ukrainian Center of Tomotherapy-Department of Chemotherapy ( Site 1451), Kropyvnytskyi, Kirovohrad Oblast
  - Sumy regional clinical oncological dispensary-Oncothoracic department ( Site 1452), Sumy, Sumska Oblast
  - Universal Clinic Oberig-Oncology Center ( Site 1461), Kyiv
- United Kingdom (6):
  - Royal Cornwall Hospitals NHS Trust ( Site 1402), Truro, Cornwall
  - University College Hospital London ( Site 1400), London, London, City of
  - Guy s & St Thomas NHS Foundation Trust ( Site 1407), London, London, City of
  - The Royal Marsden Hospital-Institute of Cancer Research ( Site 1406), London, London, City of
  - Royal Marsden NHS Foundation Trust ( Site 1408), Sutton, London, City of
  - Churchill Hospital ( Site 1404), Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trial Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26187&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 450 participants randomized, 448 received study intervention.
Period: Overall Study
Arm/Group | Pembrolizumab | Placebo
Started | 225 | 225
Treated | 224 | 224
Switchover to Pembrolizumab | 0 | 30
Retreatment With Pembrolizumab | 2 | 0
Completed | 0 | 0
Not Completed | 225 | 225
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Ongoing | 186 | 194
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Death | 34 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Placebo | Total
Number analyzed (Participants) | 225 | 225 | 450
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.3 (10.8) | 69.2 (10.7) | 69.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 82
  Male | 184 | 184 | 368
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 47 | 93
  Not Hispanic or Latino | 140 | 148 | 288
  Unknown or Not Reported | 39 | 30 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 174 | 181 | 355
  More than one race | 14 | 11 | 25
  Unknown or Not Reported | 35 | 28 | 63
Extracapsular Extension [Count of Participants; unit: Participants] — Extracapsular extension is defined as metastatic cancer extending through the nodal capsule into the peri-nodal adipose tissue. Participants were stratified by extracapsular extension (yes vs. no).
  Participants
    Yes | 89 | 98 | 187
    No | 135 | 127 | 262
    Missing Data | 1 | 0 | 1
Cortical Bone Invasion [Count of Participants; unit: Participants] — Cortical bone invasion indicates that the squamous cell carcinoma has metastasized into bone indicated by yes or no.
  Participants
    Yes | 21 | 19 | 40
    No | 203 | 206 | 409
    Missing | 1 | 0 | 1
Prior Systemic Therapy [Count of Participants; unit: Participants] — Participants were categorized as having prior systemic therapy by (yes or no).
  Participants
    Yes | 16 | 17 | 33
    No | 209 | 208 | 417

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-Free Survival (RFS) as Assessed by the Investigator and Confirmed by Biopsy
Description: RFS as assessed by investigator was defined as the time between the date of randomization to the date of first local or regional recurrence of the index lesion, distant metastasis, or death due to any cause; whichever occurred first. Participants were analyzed in the treatment group to which they were randomized. RFS as assessed by investigator is presented.
Time Frame: Up to approximately 62 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 225 | 225
Months | 53.3 [51.3 to NA] — Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 53.7 [51.8 to NA] — Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab vs Placebo; Test type: Superiority; p = 0.07243, Log Rank — One-sided p-value based on log-rank test stratified by baseline Extracapsular extension (yes versus no) and Cortical bone invasion (yes versus no) with small strata collapsed; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.53 to 1.10] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by baseline Extracapsular extension (yes versus no) and Cortical bone invasion (yes versus no) with small strata collapsed

2. Secondary Outcome: Overall Survival (OS)
Description: OS is the time from randomization to death due to any cause. Participants were analyzed in the treatment group to which they were randomized. OS is presented.
Time Frame: Up to approximately 62 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 225 | 225
Months | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.47, 95% CI 2-sided [0.87 to 2.48] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status. The change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score is presented.
Time Frame: Baseline and up to approximately 60 months
Population: All participants who had at least one dose of study intervention and one EORTC QLQ-C30 score available
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 223 | 224
Score on scale | -7.05 [-10.91 to -3.19] | -3.64 [-7.74 to 0.47]
Statistical Analysis 1: Comparison: Pembrolizumab vs Placebo; Test type: Superiority; p = 0.2227, Log Rank — Based on a cLDA model with the PRO scores as the response variable with covariates for treatment by study visit interaction, and stratification factors by Extracapsular extension, Cortical bone invasion, and Prior systemic therapy; Mean Difference (Final Values) = -3.41, 95% CI 2-sided [-8.91 to 2.09] — Based on a cLDA model with the PRO scores as the response variable with covariates for treatment by study visit interaction, and stratification factors by Extracapsular extension, Cortical bone invasion, and Prior systemic therapy

4. Secondary Outcome: Change From Baseline in Physical Functioning Using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Items 1-5 Score
Description: Change from baseline in the score of EORTC QLQ-C30 Items 1-5 is reported. The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores meant a better level of function. Participants were analyzed in the treatment group to which they were randomized. Change from baseline in EORTC QLQ-C30 physical functioning is presented.
Time Frame: Baseline and up to approximately 60 months
Population: All participants who had at least one dose of study intervention and one EORTC QLQ-C30 score available
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 223 | 224
Scores on a scale | -7.60 [-10.56 to -4.63] | -4.71 [-7.83 to -1.59]
Statistical Analysis 1: Comparison: Pembrolizumab vs Placebo; Test type: Superiority; p = 0.1874, Log Rank — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.89, 95% CI 2-sided [-7.19 to 1.42] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Percentage of Participants Who Experience an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The percentage of participants who experience at least one AE is presented.
Time Frame: Up to approximately 62 months
Population: All randomized participants who received at least one dose of study treatment
Measure: Number; unit: Percentage of participants
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 224 | 224
Percentage of participants | 94.2 | 88.8

6. Secondary Outcome: Percentage of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The percentage of participants who discontinue study treatment due to an AE is presented.
Time Frame: Up to approximately 19 months
Population: All randomized participants who received at least one dose of study treatment
Measure: Number; unit: Percentage of participants
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 224 | 224
Percentage of participants | 10.3 | 4.0

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events up to approximately 62 months.
Description: All-cause mortality included all randomized participants. Serious and other adverse events included all participants who received at least one dose of study intervention. For all-cause mortality participants were followed until they switched groups, then were followed in the crossover group. MedDRA Version: 27.0 preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to the drug are excluded.
Groups:
- Pembrolizumab (Retreatment Phase): Participants who received 400 mg pembrolizumab by intravenous (IV) infusion administered on Day 1 of each 42-day cycle (Q6W) for up to 9 cycles and experience biopsy-proven-disease recurrence received up to 18 additional cycles of pembrolizumab in an open-label design.
- Placebo Crossover: Participants who received placebo by IV infusion administered on Day 1 of each 42-day cycle (Q6W) for up to 9 cycles and experience biopsy-proven-disease recurrence may be eligible to receive up to 18 cycles of pembrolizumab 400 mg by IV infusion administered on Day 1 of each 42-day cycle (Q6W) in an open-label design.
Arm/Group | Pembrolizumab | Placebo | Pembrolizumab (Retreatment Phase) | Placebo Crossover
All-Cause Mortality (participants affected / at risk) | 34/225 | 14/225 | 1/2 | 10/30
Serious Adverse Events (participants affected / at risk) | 55/224 | 43/224 | 0/2 | 15/30
Other Adverse Events (participants affected / at risk) | 175/224 | 143/224 | 2/2 | 23/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=224) | Placebo (N=224) | Pembrolizumab (Retreatment Phase) (N=2) | Placebo Crossover (N=30)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lagophthalmos (Eye disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected seroma (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint lock (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (27) | 18 (44) | 0 (0) | 3 (3)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0) | 1 (2)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=224) | Placebo (N=224) | Pembrolizumab (Retreatment Phase) (N=2) | Placebo Crossover (N=30)
Hyperthyroidism (Endocrine disorders) | 12 (13) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 26 (26) | 12 (14) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 16 (18) | 19 (20) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 28 (41) | 28 (33) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 14 (14) | 9 (9) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (14) | 12 (13) | 1 (1) | 1 (1)
Asthenia (General disorders) | 28 (33) | 18 (19) | 0 (0) | 2 (2)
Fatigue (General disorders) | 38 (41) | 30 (31) | 0 (0) | 3 (4)
Influenza like illness (General disorders) | 7 (7) | 4 (8) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 6 (6) | 1 (1) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 6 (6) | 11 (11) | 0 (0) | 4 (4)
Influenza (Infections and infestations) | 4 (5) | 3 (3) | 0 (0) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 6 (7) | 6 (6) | 0 (0) | 2 (4)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 12 (12) | 8 (9) | 1 (1) | 3 (3)
SARS-CoV-2 test positive (Investigations) | 6 (6) | 2 (2) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 11 (11) | 10 (10) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 7 (8) | 5 (5) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (32) | 20 (23) | 0 (0) | 3 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (14) | 8 (9) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (10) | 5 (6) | 0 (0) | 2 (2)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (12) | 18 (40) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 4 (7) | 0 (0) | 2 (3)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (24) | 17 (19) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 9 (9) | 9 (11) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 5 (5) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 19 (21) | 16 (17) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 6 (6) | 3 (4) | 0 (0) | 2 (2)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 7 (7) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 0 (0) | 2 (3)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 19 (24) | 27 (40) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 42 (50) | 18 (20) | 0 (0) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 20 (26) | 17 (17) | 0 (0) | 2 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (13) | 5 (5) | 0 (0) | 3 (7)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (15) | 12 (19) | 0 (0) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors (ICMJE) authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT03833167/Prot_SAP_000.pdf